CLINICAL TRIAL: NCT02039206
Title: The Influence of Deep Repetitive Transcranial Magnetic Stimulation (TMS) on Cerebellar Signs in Patients With Spinocerebellar Ataxia Type 3 (SCA3 - Machado Joseph Disease)
Brief Title: The Influence of Deep TMS on Cerebellar Signs in Patients With Machado Joseph Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brainsway (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MJD MEIR dTMS; 0059-13-MMC (Other: BRAINSWAY)
Record Dates: First submitted 2013-12-29; First posted 2014-01-17 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Machado Joseph Disease (SCA3)
Keywords: Machado Joseph disease; Deep TMS; TMS; Transcranial Magnetic Stimulation; SCA3; Magnetic Stimulation; Brainsway
MeSH Terms: conditions — Machado-Joseph Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Deep TMS
  Interventions: Device: Deep TMS

INTERVENTIONS:
Device: Deep TMS — 1Hz Stimulation

SUMMARY:
To test the effects of low frequency deep rTMS using the novel HCERMJD-coil on cerebellar deficits in patients with SCA3 and to establish its safety in this population.

Investigator is anticipate that stimulation of the cerebellum with the novel HCERMJD-coil may induce significantly therapeutic effects in patients with SCA3 and will pave the way for establishing a novel and effective treatment for this disorder.

ELIGIBILITY:
Inclusion Criteria:

* SCA3 patients aged 20 - 80 years, with detectable clinical signs and confirmed genetic diagnosis.

Exclusion Criteria:

1. Patients who have concomitant epilepsy.
2. History of seizure or heat convulsion.
3. Patients on neuroleptics.
4. Patients with dementia (MMSE<25) or any unstable medical disorder.
5. History or current unstable hypertension.
6. History of head injury or neurosurgical interventions.
7. History of any metal in the head (outside the mouth).
8. Known history of any metallic particles in the eye, implanted cardiac pacemaker, implanted neurostimulators, surgical clips (above the shoulder line) or any medical pumps.
9. History of frequent or severe headaches.
10. History of migraine.
11. History of hearing loss.
12. History of cochlear implants
13. History of drug abuse or alcoholism.
14. Pregnancy or not using a reliable method of birth control.
15. Participation in current clinical study or clinical study within 30 days prior to this study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Scale for the Assessment and Rating of Ataxia (SARA) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Gordon, Prof., Principal Investigator — Meir Health Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel